CLINICAL TRIAL: NCT01720394
Title: Efficacy of Induction of Labor on Term Using a Double Balloon Catheter Compared to Dinoprostone Vaginal-insert - a Multicenter Randomized Controlled Trial
Brief Title: Efficacy of Induction of Labor on Term Using a Double Balloon Catheter Compared to Dinoprostone Vaginal-insert
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other); Medical University Innsbruck (Other); Klinikum Klagenfurt am Wörthersee (Other); University of Salzburg (Other); Hospital Hartberg, Austria (Unknown); Hospital Braunau, Austria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUG-CRB-2012
Record Dates: First submitted 2012-06-25; First posted 2012-11-02 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Cervical Ripening; Induction of Labor
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical ripening balloon (Experimental): primary treatment with the cervical ripening balloon on day 1. removal of the balloon latest after 12 h. If no progression of labor (Bishop Score ≥ 9 and/or cervical opening ≥ 3 cm) continuing of standard treatment using dinoprostone vaginal-inserts on day 2 and if necessary on day 3.
  Interventions: Device: Cervical Ripening Balloon, Cook Medical Inc.
- Propess (Active Comparator): Primary treatment using dinoprostone-vaginal-inserts on day 1-3 if no progression of labor (Bishop Score ≥ 9 and/or cervical dilatation ≥ 3 cm)
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Device: Cervical Ripening Balloon, Cook Medical Inc. — Application of the cervical ripening double-balloon (filled with 2x 80ml) on day 1.
  Other Names: Cook cervical ripening balloon, Cook OB/GYN, Spencer, IN, 47460 USA - CE 0088, 400470E; Propess-vaginal-insert (Dinoprostone 10mg), Ferring Arzneimittel Ges.m.b.H., 1100 Vienna, Austria
  Arms: Cervical ripening balloon
Drug: Dinoprostone — Application of Propess-vaginal-insert, (Dinoprostone 10mg - Ferring Arzneimittel Ges.m.b.H., 1100 Vienna, Austria) for labor induction on day 1-3 in therapy arm 2.
  Other Names: Propess, (Dinoprostone 10mg), Ferring Arzneimittel Ges.m.b.H., 1100 Vienna, Austria
  Arms: Propess

SUMMARY:
The purpose of the study is to determine the efficacy of a silicone-double-balloon-catheter for cervical ripening and labor induction in women with unfavorable cervix (Bishop Score not greater than 6) compared to medical treatment using a dinoprostone slow-release-vaginal-insert.

ELIGIBILITY:
Inclusion Criteria:

* medical indication for induction of labor
* 18 years of age
* signed informed consent
* cephalic presentation
* no PROM
* 37+0 - 42+0 weeks of gestation
* Bishop-Score ≤ 6
* no contra-indication for medical induction of labor
* no clinical signs of infection

Exclusion Criteria:

* fetal anomalies
* contra-indications for medical induction of labor
* placental pathologies
* St.p. surgery with opening the uterine cavity (incl. caesarean section)
* PROM
* multiple gestations
* < 37-0 weeks of gestation
* St.p. cervical tear

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2013-11; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
time interval from primary treatment to delivery | maximum of 72 hours
  the time interval between the first application of the cervical ripening balloon (therapy arm 1) to delivery and the time between first application of dinoprostone vaginal-insert (therapy arm 2) to delivery is measured

SECONDARY OUTCOMES:
progress of labor | maximum of 72 hours
  time from balloon-application to dilatation of the cervix (cervical opening > 3cm, or Bishop Score ≥ 9 ) in therapy arm 1 and from dinoprostone-vaginal-insert-application to dilatation of the cervix (cervical opening > 3cm, or Bishop Score ≥ 9 ) in therapy arm 2
vaginal delivery | maximum of 72 hours
  Number of patients who achieve spontaneous vaginal delivery or vaginal-operative delivery in therapy arm 1 and 2.
failed induction of labor | maximum of 72 hours
  Number of patients who received caesarean section after frustrating induction of labor. Frustrating induction is defined as application of the cervical-ripening-balloon + 2 times application of dinoprostone-vaginal-insert in therapy arm 1 and 3 times application of dinoprostone-vaginal-insert in therapy arm 2.
patient's satisfaction | participants will be followed for the duration of hospital stay, an expected average of 5-7 days
  Patient's satisfaction with treatment is evaluated with a questionnaire within 48 h after delivery
maternal parameters | primary treatment - 48h postpartal, leading to a maximum time frame of 5 days
  signs of infection (temperature, CRP, WBC), childbirth--related injuries,need for epidural in therapy arm 1 and 2.
fetal parameters | primary treatment - fetal hospital discharge, with an expected maximum of 3 months
  umbilical cord blood values, apgar score, fetal birth weight,number of admissions to ICU and days at ICU in therapy arm 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Klaritsch, MD, Study Chair — Medical University of Graz; Philipp Reif, MD, Principal Investigator — Medical University of Graz
Locations (7):
- Austria (7):
  - Abteilung für Gynäkologie und Geburtshilfe, Krankenhaus St. Josef Braunau, Braunau am Inn
  - Universitätsklinik für Frauenheilkunde und Geburtshilfe, Medizinische Universität Graz, Graz
  - Abteilung für Gynäkologie und Geburtshilfe, LKH Hartberg, Hartberg
  - Universitätsfrauenklinik Innsbruck, Medizinische Universität Innsbruck, Innsbruck
  - Abteilung für Gynäkologie und Geburtshilfe, Perinatalzentrum, Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Universitätsklinik für Frauenheilkunde und Geburtshilfe, Landeskrankenhaus Salzburg - Universitätsklinikum der Paracelsus Medizinischen Privatuniversität, Salzburg
  - Universitätsfrauenklinik Wien, Abteilung für Geburtshilfe und fetomaternale Medizin, Medizinische Universität Wien, Vienna

REFERENCES:
- [Background] Martin JA, Hamilton BE, Sutton PD, Ventura SJ, Menacker F, Kirmeyer S. Births: final data for 2004. Natl Vital Stat Rep. 2006 Sep 29;55(1):1-101. PMID 17051727
- [Background] Sherman DJ, Frenkel E, Tovbin J, Arieli S, Caspi E, Bukovsky I. Ripening of the unfavorable cervix with extraamniotic catheter balloon: clinical experience and review. Obstet Gynecol Surv. 1996 Oct;51(10):621-7. doi: 10.1097/00006254-199610000-00022. PMID 8888040
- [Background] Husslein P. Use of prostaglandins for induction of labor. Semin Perinatol. 1991 Apr;15(2):173-81. No abstract available. PMID 1876873
- [Background] Boulvain M, Kelly A, Lohse C, Stan C, Irion O. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2001;(4):CD001233. doi: 10.1002/14651858.CD001233. PMID 11687101
- [Background] Prager M, Eneroth-Grimfors E, Edlund M, Marions L. A randomised controlled trial of intravaginal dinoprostone, intravaginal misoprostol and transcervical balloon catheter for labour induction. BJOG. 2008 Oct;115(11):1443-50. doi: 10.1111/j.1471-0528.2008.01843.x. Epub 2008 Aug 19. PMID 18715244
- [Background] Kehl S, Ehard A, Berlit S, Spaich S, Sutterlin M, Siemer J. Combination of misoprostol and mechanical dilation for induction of labour: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2011 Dec;159(2):315-9. doi: 10.1016/j.ejogrb.2011.09.010. Epub 2011 Oct 2. PMID 21962943
- [Background] Pennell CE, Henderson JJ, O'Neill MJ, McChlery S, Doherty DA, Dickinson JE. Induction of labour in nulliparous women with an unfavourable cervix: a randomised controlled trial comparing double and single balloon catheters and PGE2 gel. BJOG. 2009 Oct;116(11):1443-52. doi: 10.1111/j.1471-0528.2009.02279.x. Epub 2009 Jul 28. PMID 19656148
- [Background] Mei-Dan E, Walfisch A, Suarez-Easton S, Hallak M. Comparison of two mechanical devices for cervical ripening: a prospective quasi-randomized trial. J Matern Fetal Neonatal Med. 2012 Jun;25(6):723-7. doi: 10.3109/14767058.2011.591459. Epub 2011 Aug 2. PMID 21806490
- [Background] Calder AA. Review of prostaglandin use in labour induction. Br J Obstet Gynaecol. 1997 Oct;104 Suppl 15:2-7; discussion 20-5. No abstract available. PMID 9366720
- [Background] Cromi A, Ghezzi F, Uccella S, Agosti M, Serati M, Marchitelli G, Bolis P. A randomized trial of preinduction cervical ripening: dinoprostone vaginal insert versus double-balloon catheter. Am J Obstet Gynecol. 2012 Aug;207(2):125.e1-7. doi: 10.1016/j.ajog.2012.05.020. Epub 2012 Jun 1. PMID 22704766
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- See also: Drug Information on Dinoprostone — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0000363246&QV1=DINOPROSTONE